CLINICAL TRIAL: NCT00676390
Title: Estimated Physical Activity of Congestive Heart Failure Patients by a Physical Activity Questionnaire : Concordance Study.
Brief Title: Estimated Physical Activity of Congestive Heart Failure Patients by a Physical Activity Questionnaire
Acronym: H2OBis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0708046; 2007- A00615-48 (Other: AFSSAPS); DGS 2007-0434 (Other: DGS)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Congestive Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Congestive Heart failure patients
  Interventions: Other: doubly labelled water and questionnaire

INTERVENTIONS:
Other: doubly labelled water and questionnaire — 0.075 g.kg-1 and 2H2O et 0.15 g.kg-1 de H218O per oral at inclusion visit. physical activity questionnaire at inclusion visit

SUMMARY:
The treatment and follow-up of congestive heart failure (CHF) represents a major part of France's health expenses. The beneficial effects of cardiac rehabilitation is well established, especially regarding the reduction of dyspnea, exercise limitation and fatigue and leads ultimately to a better quality of life. Maintaining these benefits in secondary prevention requires an improvement in daily physical activity, which is challenging and supposes a close follow-up difficult to perform on a daily living basis. However, a better knowledge of the type and dose of daily physical activity of this population would be very beneficial for the practitioner to prescribe or advise individually the type and the dose of physical activity required to maintain the benefits of cardiac rehabilitation. To date, only a physical activity questionnaire adapted to CHF could provide information regarding both the type and dose of daily physical activity. Such a questionnaire has been developed by our research team and allows an estimation of daily energy expenditure as well as the daily energy expended in its physical activity dimensions (rest, activities < 3 MET, activities between 3 and 5 MET, and activities > 5 MET). During its first step of validation, daily and physical activity energy expenditure estimated by this questionnaire was correlated to various factors of physical condition and notably, to peak V'O2 (R=0.71), prognostic factor largely recognized in CHF. A second step of validation was a pilot study comparing the estimation of daily energy expenditure by the questionnaire with a measurement of free-living daily energy expenditure with the doubly labelled water (DLW) method in 11 middle-aged males patients suffering CHF (NYHA I to III). Daily energy expenditure estimated from the questionnaire was very close to daily energy expenditure measured from the DLW method (R2 = 0.81; individual relative error < 7%). However, the high cost of the DLW method reduced the population studied to a small sample, which is a major limitation of this study since the sample was somewhat different to general CHF population in France.

DETAILED DESCRIPTION:
Therefore, the aim of the present study was to assess the validity of the questionnaire against the DLW method in a larger population of 30 patients with CHF more representative of the general population with CHF, including men and women, NYHA I to IV, with a larger age panel. Along with this concordance study, a measurement of the energy cost of specific physical activities of daily life is performed with an ambulatory gaz analyzer method to further validate the calculation method of daily energy expenditure from the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Congestive Heart Failure
* Stade II, III of NYHA
* Between 20 to 80 years old
* EF < 45%
* Written informed consent
* French language

Exclusion Criteria:

* Corticotherapy
* Thyroid dysfunction
* Cachectic status

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To validate a physical activity questionnaire adapted to congestive heart failure patients by the questionnaire comparing with a measurement of free-living daily energy expenditure with the doubly labelled water. | D14 visit

SECONDARY OUTCOMES:
To determinate the energy cost of specific physical activities of daily life performed with an ambulatory gaz analyzer method | D14 visit

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ROCHE, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Service de Physiologie Clinique et de l'Exercice, CHU de Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Background] Garet M, Barthelemy JC, Degache F, Costes F, Da-Costa A, Isaaz K, Lacour JR, Roche F. A questionnaire-based assessment of daily physical activity in heart failure. Eur J Heart Fail. 2004 Aug;6(5):577-84. doi: 10.1016/j.ejheart.2003.11.022. PMID 15302005